CLINICAL TRIAL: NCT07293884
Title: Efficacy of Nebulized Versus Intravenous N- Acetylcysteine in Airway Clearance in Broncheictasis
Brief Title: N- Acetylcysteine in Airway Clearance in Broncheictasis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sahar Refaat Mahmoud, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NAcetylcysteine broncheictasis
Record Dates: First submitted 2025-11-26; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Broncheictasis
Keywords: broncheictasis; N-acetylecysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV N Acetyle cysteine (Active Comparator): Intervention: N Acetyle cysteine given by IV injection
  Interventions: Drug: N Acetyle cysteine given by IV injection
- Nebulized N Acetyle cysteine (Active Comparator): Intervention: Nebulized N Acetyle cysteine
  Interventions: Drug: Nebulized N Acetyle cysteine

INTERVENTIONS:
Drug: N Acetyle cysteine given by IV injection — Arm: IV N Acetyle cysteine
  Arms: IV N Acetyle cysteine
Drug: Nebulized N Acetyle cysteine — Arm: Nebulized N Acetyle cysteine
  Arms: Nebulized N Acetyle cysteine

SUMMARY:
It has been deduced that reducing the production of mucus or improving the clearance of sputum in the airway is the key to enhance the therapeutic efficacy for bronchiectasis . Mucoactive drugs are commonly used to clear the airway in mucus hypersecretion diseases. Currently, investigators have found that N-acetylcysteine (NAC), an effective mucolytic agent, not only reduces the viscosity and elasticity of sputum, but it also has anti-inflammatory and antioxidant activity.

Additionally, the Spanish guidelines on the treatment of bronchiectasis indicate that the use of N-acetylcysteine should be considered for patients with bronchiectasis and COPD. Therefore, as a classic mucolytic agent with antioxidant and anti-inflammatory properties, N-acetylcysteine can be effective in the treatment of bronchiectasis

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged above 18 years old; with a diagnosis of bronchiectasis who are admitted to chest department due to acute exacerbation

Exclusion Criteria:

* current smokers, a known allergy to N-acetylcysteine; pregnancy or lactation (for women); primary diagnosis of COPD or asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
sputum viscosity score | At the end of 1 week of treatment
  Sputum viscosity score \(0\): Normal (liquid)\(1\): Mildly increased viscosity (fluid)\(2\): Moderately increased viscosity (viscous)\(3\): Severely increased viscosity (sticky)
Amount of sputum | At the end of 1 week treatment
Expectoration difficulty score | At the end of 1 week of treatment
  Expectoration difficulty score \(0\): No difficulty\(1\): Mild difficulty\(2\): Moderate difficulty\(3\): Marked difficulty

SECONDARY OUTCOMES:
Need for mechanical ventilation | At the end of 1 week of treatment

IPD SHARING:
Plan to Share IPD: Undecided